CLINICAL TRIAL: NCT03399019
Title: Usefulness of Bispectal Index (BIS) on Depth of Sedation With Dexmedetomidine, Propofol and Midazolam During Spinal Anesthesia : a Prospective Randomized Study
Brief Title: Bispectral Index(BIS) on Depth of Sedation With Dexmedetomidine, Propofol and Midazolam During Spinal Anesthesia
Acronym: BIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2016-I097
Record Dates: First submitted 2017-01-02; First posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Sedation; Anesthesia, Spinal
Keywords: Bispectral index monitor
MeSH Terms: interventions — Dexmedetomidine; Propofol; Midazolam

STUDY DESIGN:
Intervention Model Description: This study compares to the same intervention (monitor BIS scores and OAA/S scores timely) between all of three sedative drugs.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dexmedetomidine (Experimental): Dexmedetomidine
  : initial loading 0.5- 1 mng/kg for 10 minutes and maintenance 0.2-0.7mng/kg/hr
  Check BIS (bispectral index) score and OAA/S (Observer assessment of alertness/sedation score) by time
  Interventions: Drug: Dexmedetomidine
- Propofol (Active Comparator): Propofol
  : 0.75-3 mg/kr/hr continous infusion Check BIS (bispectral index) score and OAA/S (Observer assessment of alertness/sedation score) by time
  Interventions: Drug: Propofol
- Midazolam (Active Comparator): Midazolam
  : initial loading 0.5- 1 mng/kg for 10 minutes and maintenance 0.2-0.7mng/kg/hr
  Check BIS (bispectral index) score and OAA/S (Observer assessment of alertness/sedation score) by time
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — initial loading dose (0.5 ~ 1㎍/kg for 10 minutes) and maintenance infusion (0.2-0.7㎍/kg/hr)
  Arms: Dexmedetomidine
Drug: Propofol — continuous infusion (0.75-3mg/kg/hr)
  Arms: Propofol
Drug: Midazolam — 0.05mg/kg bolus injection and if not OAA/S ≤ 3 within 5 minutes, add 0.01mg/kg at intervals of 1~2 minutes
  Arms: Midazolam

SUMMARY:
This study is to investigate on the objective relevance between bispectral index (BIS) and Observer's assessment of alertness/sedation (OAA/S) scale in patients sedated with Midazolam, propofol and dexmedetomidine during spinal anesthesia. Also, we will evaluate the reflection of actual sedation levels on BIS monitoring.

DETAILED DESCRIPTION:
Sedation is an important element of regional anesthesia during surgery, which allows to finish surgery smoothly by reducing patients' anxiety and fear who undergo regional and local anesthesia.

If adequate sedation is not maintained during regional anesthesia, surgery may be disturbed by patient's movement. This can cause the patient to be physically and mentally stressed with discomfort.

Commonly used measurement to determine the adequate sedation level relies on subjective physician's assessment such as scoring for response to talk, shake and pain. This measurement is unreliable and not continuous.

Recently, BIS is used to guide sedation during spinal anesthesia as an objective monitoring method in many studies. but previous studies result contrasting in the correlation between BIS and sedation levels with lack in evaluation between sedative drugs.

In this study, the investigators will investigate the usefullness of BIS monitoring during regional anesthesia with sedation and evaluate the suitability of correlation BIS and OAA/S between drugs (midazolam, propofol and dexmedetomidine). The anesthetic and sedation protocol will be standardized.

ELIGIBILITY:
Inclusion Criteria:

* Patients who scheduled for knee arthroscopic surgery under spinal anesthesia

Exclusion Criteria:

* Patients with a history of hepatic, renal, cardiovascular disease, and those who have allergy to study drugs (dexmedetomidine, propofol, midazolam).
* Hemodynamically unstable patients.
* Patients who is noncommunicative.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-09-05 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
correlation between BIS and OAA/S (observer's assessment of alertness/sedation) score | 1 day
  Statistically significant (p<0.05) correlations between BIS (range of 0-100) and OAA/S scale (range of 1-5) in dexmedetomidine, propofol and midazolam.

SECONDARY OUTCOMES:
The amount of rescue analgesics (fentanyl in mg) and rescue hypnotic (propofol in mg) | 1 day
  The amount of rescue hypnotics due to insufficient sedation (total additional volume of propofol in mg) and rescue analgesics (total additional volume of fentanyl in mng) due to insufficient pain control

CONTACTS AND LOCATIONS:
Overall Officials: Soo Kyung Lee, M.D, Study Director — Hallym University Medical Center
Locations (1):
- Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kato T, Koitabashi T, Ouchi T, Serita R. The utility of bispectral index monitoring for sedated patients treated with low-dose remifentanil. J Clin Monit Comput. 2012 Dec;26(6):459-63. doi: 10.1007/s10877-012-9379-4. Epub 2012 Jul 25. PMID 22828857
- [Background] Venn RM, Grounds RM. Comparison between dexmedetomidine and propofol for sedation in the intensive care unit: patient and clinician perceptions. Br J Anaesth. 2001 Nov;87(5):684-90. doi: 10.1093/bja/87.5.684. PMID 11878517
- [Background] Kasuya Y, Govinda R, Rauch S, Mascha EJ, Sessler DI, Turan A. The correlation between bispectral index and observational sedation scale in volunteers sedated with dexmedetomidine and propofol. Anesth Analg. 2009 Dec;109(6):1811-5. doi: 10.1213/ANE.0b013e3181c04e58. PMID 19923507